CLINICAL TRIAL: NCT03227367
Title: Platelet Rich Fibrin/Biphasic Calcium Phosphate Impairs Osteoclasts Differentiation and Promotes Apoptosis by the Intrinsic Mitochondrial Pathway in Chronic Periodontitis
Brief Title: Osteoclast Impairment in Chronic Periodontitis by Regenerative Materials.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Director post graduate studies, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MU-107-IEC/2014
Record Dates: First submitted 2017-06-25; First posted 2017-07-24 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Periodontal Disease; Periodontal Bone Loss; Osteoclastic Bone Loss
Keywords: biomaterials; apoptosis; bone regeneration
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Control group: (Healthy individuals) comprised of 25 participants with clinically healthy periodontium.
  Test group: (Chronic periodontitis patients) comprised of 25 participants with signs of clinical inflammation and bone loss.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Mononuclear cells isolated from the peripheral blood of 25 chronic periodontitis patients were interveened with 1ml/well preparation of Platelet rich fibrin(PRF), Biphasic calcium phosphate (BCP) and PRF and BCP combination in-vitro.
  Interventions: Other: other : PRF
- control group (Other): Mononuclear cells isolated from the peripheral blood of healthy individuals in-vitro.
  Interventions: Other: other : PRF

INTERVENTIONS:
Other: other : PRF — mononuclear cells from the peripheral blood of chronic periodontitis patients were intervened with PRF, BCP and PRF/BCP combination
  Other Names: others : BCP; others : PRF/BCP combination

SUMMARY:
The present study is an effort to investigate the hypothesis that Platelet Rich Fibrin/Biphasic Calcium Phosphate may play a role in inhibiting osteoclasts differentiation and in bone loss.

DETAILED DESCRIPTION:
Study design

Fifty-five individuals from a suburban population were recruited. Out of them, 5 individuals refused to participate in the study. Finally, 50 participants were selected and divided into two groups, control group [Healthy individuals]: 25 Males/Females, aged 25 to 35 years and test group [Chronic periodontitis patients]: 25 Males/Females aged 30 to 45 years.

Demographic variables and periodontal parameters were measured in both the groups.The investigators explored the effect of Platelet rich fibrin (PRF)/Biphasic calcium phosphate (BCP) on differentiation and survival of osteoclasts obtained from peripheral blood of Chronic Periodontitis patients.

ELIGIBILITY:
Inclusion criteria: (Control group)

* Subjects with age group between 30 to 45 years.
* Non-smokers.
* No previous history of periodontal treatment.

Inclusion Criteria: (Test group)

* Subjects with age group between 30 to 45 years.
* Presence of atleast 20 teeth
* More than 30% of the sites with clinical attachment loss.
* Non-smokers.
* No previous history of periodontal treatment.

Exclusion Criteria: ( both the groups)

* Individuals with systemic disease
* Subjects under antibiotics or anti-inflammatory drugs within the previous 3 months.
* Pregnant and lactating women.
* Allergic to antibiotics.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2017-03-18 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | base line
  probing pocket dept was measured using Williams periodontal probe at base line

SECONDARY OUTCOMES:
Protein expression on osteoclast cells was estimated with BCP, PRF alone and BCP/PRF combination. | 24 hours from baseline
  Protein expression on cells was analyzed using Western blot in all the groups
The activity of caspase-3 in OCs. | 24 hours from base line
  The activity of caspase-3 was seen in OCs in all the groups

CONTACTS AND LOCATIONS:
Overall Officials: shila samuel, MS, PhD, Principal Investigator — VRR diagnostic institute chennai; jaideep mahendra, MDS,PhD, Principal Investigator — meenakshi ammal dental college chennai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu CL, Lee SS, Tsai CH, Lu KH, Zhao JH, Chang YC. Platelet-rich fibrin increases cell attachment, proliferation and collagen-related protein expression of human osteoblasts. Aust Dent J. 2012 Jun;57(2):207-12. doi: 10.1111/j.1834-7819.2012.01686.x. PMID 22624763
- [Result] Colucci S, Mori G, Brunetti G, Coricciati M, Pignataro P, Oranger A, Cirulli N, Mastrangelo F, Grassi FR, Grano M. Interleukin-7 production by B lymphocytes affects the T cell-dependent osteoclast formation in an in vitro model derived from human periodontitis patients. Int J Immunopathol Pharmacol. 2005 Jul-Sep;18(3 Suppl):13-9. PMID 16848983